CLINICAL TRIAL: NCT04650256
Title: Application of Chinese Herbal Complementary and Alternative Medicine (CAM) to Improve Human Health and to Further Botanical and Horticultural Sciences
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: VAUGHN-JORDAN FOUNDATION, INC. (Unknown); Florida Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Hu, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200491
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Skin Toxicity
Keywords: Breast cancer; Radiotherapy; Complementary and alternative medicine
MeSH Terms: conditions — Breast Neoplasms | interventions — Complementary Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAM arm (Experimental): Participants will be given the CAM intervention during scheduled, standard of care radiotherapy (up to 6 weeks) and 8-12 weeks (weeks 14-18) after radiotherapy.
  Interventions: Other: Complementary and alternative medicine (CAM)

INTERVENTIONS:
Other: Complementary and alternative medicine (CAM) — CAM will be applied topically on the chest wall once during the day (or immediately after radiotherapy) and once at night daily.

SUMMARY:
The purpose of this research is to study a Chinese herbal Complementary and Alternative Medicine (CAM) product for the temporary relief of pain and itching after radiotherapy (RT). This is an over-the-counter product with 1% menthol as an active ingredient.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with newly diagnosed breast carcinoma
* > 18 years of age
* Post-mastectomy with or without reconstruction
* Stage II-IIIb with any receptor status
* All races and ethnicities are eligible
* Patients must be able to consent in English or Spanish
* Plan to receive adjuvant radiotherapy to the chest wall +/- regional lymph nodes
* RT will involve standard fractionation use of 3D conformal or Intensity-modulated RT (IMRT)
* Willing to sign protocol consent form
* Patients are allowed to receive adjuvant hormonal therapy and/or targeted therapies such as trastuzumab prior to, during and/or after radiation therapy.
* Patients may receive chemotherapy before or after radiation therapy

Exclusion Criteria:

* Prior radiation to the involved breast or chest wall
* Concurrent chemotherapy
* Unable or unwilling to sign informed consent
* Unable to speak English or Spanish
* Pregnant women
* Clinical or pathologic stage T4
* Metastatic disease
* Connective tissue disorder including Systemic Lupus Erythematosus and Scleroderma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients free of clinically relevant skin toxicities | Up to 18 weeks.
  Clinically relevant skin toxicities - Grade 2 with moist desquamation or Grade 3 or higher using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) as evaluated by the treating clinician.

SECONDARY OUTCOMES:
SD-16 scores | Up to 18 weeks.
  Skindex 16 (SD-16) will be used to assess patients' self-assessment of skin effects. SD-16 has a total score ranging from 0-96 with a higher score indicating greater skin effects.
Functional Assessment of Cancer Therapy-Breast (FACT-B) scores | Up to 18 weeks.
  FACT-B in breast cancer patients will be used to obtain patient's self-assessment of health-related quality of life. FACT-B has a total score ranging from 0-148 with a higher score indicating a better quality of life.
High-sensitivity C-reactive protein (hsCRP) values | Up to 6 weeks
  The inflammatory biomarker, plasma high-sensitivity C-reactive protein (hsCRP) will be evaluated using blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Hu, PhD, Principal Investigator — U. of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No